CLINICAL TRIAL: NCT00642928
Title: Randomized, Dose-finding Study of BF 2.649 5, 10 20 and 40 mg/d in Comparison to Placebo in Excessive Daytime Sleepiness in Parkinson's Disease Patients (PD)
Brief Title: Dose Range Finding Study of BF2.649 Versus Placebo to Treat Excessive Daytime Sleepiness in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07-02 / BF 2.649; 2007-003512-57 (EudraCT Number)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Excessive Daytime Sleepiness; Parkinson's Disease
Keywords: Excessive Daytime Sleepiness; Parkinson's disease
MeSH Terms: conditions — Disorders of Excessive Somnolence; Parkinson Disease | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BF 2.649-5 mg (Experimental)
  Interventions: Drug: BF 2.649 5 mg
- BF 2.649 10 mg (Experimental)
  Interventions: Drug: BF 2.649 10 mg
- BF 2.649 20 mg (Experimental)
  Interventions: Drug: BF 2.649 20 mg
- BF 2.649 40 mg (Experimental)
  Interventions: Drug: BF 2.649 40 mg

INTERVENTIONS:
Drug: Placebo — 1 capsule per day during 4 weeks
  Arms: Placebo
Drug: BF 2.649 5 mg — one BF 2.649 capsule of 5 mg per day during 4 weeks
  Other Names: pitolisant
  Arms: BF 2.649-5 mg
Drug: BF 2.649 10 mg — One BF 2.649 capsule of 10 mg per day during 4 weeks
  Other Names: pitolisant
  Arms: BF 2.649 10 mg
Drug: BF 2.649 20 mg — One BF 2.649 capsule of 20 mg per day during 4 weeks
  Other Names: pitolisant
  Arms: BF 2.649 20 mg
Drug: BF 2.649 40 mg — One BF 2.649 capsule of 40 mg per day during 4 weeks
  Other Names: pitolisant
  Arms: BF 2.649 40 mg

SUMMARY:
The objective of this trial is to define the minimum effective dose of BF 2.649 between 5 mg, 10 mg, 20 mg or 40 mg versus placebo in reducing the Excessive Daytime Sleepiness of Parkinson's disease patients

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by resting tremor, rigidity, bradykinesia and loss of postural reflexes that affects 1% of the North American population. Besides these motor problems there are also so called non-motor problems.

Excessive daytime sleepiness (EDS) is a bothersome non-motor problem, which affects 20% to 50% of all PD patients and currently, there isn't any registered treatment for that trouble.

The study medication BF2.649 tested here is a novel, highly potent, selective, orally active inverse agonist at the histamine H3 receptor, therefore strengthens histaminergic transmission in the brain and increases wakefulness EDS is characterized by daytime somnolence and sudden sleep episodes. This problem has several consequences, e.g., an impairment of quality of life, an interference with activities of daily living and other handicaps in the management of social and family affairs.

The primary endpoint of this study will be measured by the change in the well-validated Epworth sleepiness scale (ESS). The ESS is a simple self-administered 8-item questionnaire. The outcome is to get an impression about the level of the daytime sleepiness in several real-life situations.

On the basis of this pharmacological and clinical rationale it is considered relevant to carry out a dose-finding study for this original, non-amphetamine molecule in PD patients affected by excessive daytime sleepiness. PD severity will be assessed by the routinely used UPDRS.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic Parkinson disease

* Hoehn and Yahr < 5
* Stable treatment of Parkinson disease for at least 4 weeks
* Excessive Daytime Sleepiness : Epworth scale superior or equal to 13
* None psychostimulant treatment intake for 2 weeks

Exclusion Criteria:

* Other degenerative parkinsonian syndrome
* other condition than PD that is the primary cause of excessive daytime sleepiness
* Severe depression or suicidal risk
* Pregnant or breast-feeding women
* Patients having an occupation that requires night shift
* History of drugs, alcohol, narcotic or other substance abuse or dependence
* Refusal from the patient to stop any current therapy for excessive daytime sleepiness or predictable risks for the patient to stop the therapy
* Any significant abnormality in the physical examination or clinical laboratory results e.g. liver or kidney function deficiency
* Any significant serious abnormality of the ECG e.g. myocardial infarction,
* Electrocardiogram corrected QT interval higher than 450 ms
* Other active clinically significant illness which could interfere with the study conduct or contra-indicate the study treatments or put patients at risk
* Dementia with MMS inferior or equal to 24
* Patients taking associated treatments which are not allowed during the study course and which cannot be stopped before the inclusion visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale scores (ESS) | At selection visit (Day-14 to Day-7)/Inclusion visit (Day0)/ Interim visit (Day14)/Final visit (Day28)

SECONDARY OUTCOMES:
Mean number of daytime sleep or sleepiness episodes and their duration | During 5 days before each visit
frequency of sleep attacks | recorded at each visit
UPDRS III for motor function | at each visit
Clinical global impression scale | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: ARNULF Isabelle, Principal Investigator — Pitié-Salpêtrière Hospital, Paris, France; Carsten Moeller, Principal Investigator — Universitätsklinikum Giessen und Marburg, Marburg, Germany
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France